CLINICAL TRIAL: NCT03099941
Title: The Comparison of the Effects of Two Different Feedback in the Core Stabilization Training for Patients With Chronic Nonspecific Low Back Pain (CNLBP): Randomized Parallel Group Trial
Brief Title: The Effectiveness of Two Different Feedbacks in Core Stabilization Education for Chronic Nonspecific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, GÜLVİN DİLAN CANAN, Director Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IstanbulFizyoterapi
Record Dates: First submitted 2017-03-21; First posted 2017-04-04 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Low Back Pain, Mechanical, Biofeedback, Pain, Chronic
Keywords: Low Back Pain, Mechanical, Biofeedback, Pain, Chronic
MeSH Terms: conditions — Low Back Pain; Pain; Bronchiolitis Obliterans Syndrome | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofeedback group (Experimental): The biofeedback application which helps patient to understand neutral position and how to maintain it in exercises that are prescribed by the physical therapist
  Interventions: Other: Biofeedback
- Physical therapist feedback group (Active Comparator): In physical therapist feedback group feedback applied by oral and tactile stimulation of physical therapist to helps patient to understand neutral position and how to maintain it in exercises that are prescribed
  Interventions: Other: Biofeedback

INTERVENTIONS:
Other: Biofeedback — The aim of this study is to investigate effects of a biofeedback application that is alternative to physical therapist feedback in core stabilization training of patients with CNLBP.

SUMMARY:
Abstract. Insufficient motor control mechanism of transversus abdominus and multifidus muscles is the most important cause of the chronic nonspecific low back pain (CNLBP). Recently, applications sre developed that generates audio and vibrant stimuli in response to anteroposterior and mediolateral rotations and can be adapted according to subject-specific movement sensitivity.

Objective. The objective of this study was to compare effects of a biofeedback application that is alternative to physiotherapist feedback in core stabilization training of patients with chronic nonspecific low back pain.

Design. This study was a parallel group randomized controlled trial with outcome assessment.

Patients. The participants were 38 patients with chronic (≥12 weeks) nonspecific low back pain.

Interventions. Patients were randomly assigned to receive either physiotherapist feedback or Perfect Practice (Level Belt Pro Inc.) biofeedback. Patients in both groups received 12 sessions, 30 minutes of three weekly graded functional core education trial.

Measurements. Primary outcome measures were muscle strength (transversus abdominus and multifidus) pain intensity (Visual Analog Scale) and functional level (Revised Oswestry Disability Index); secondary outcomes were flexibility (modified Schober test), range of motion (universal goniometer), proprioception (Active Reposition Test), patient beliefs (Fear Avoidance Beliefs Questionnaire), psychological status (Beck Depression Index), and quality of life(36 Item Short-Form Health Survey questionnaire [SF-36]).

Limitations. Outcome measures for muscle strength did not include objective assesment.

Keywords. Chronic low back, core stabilization training, biofeedback, pain, function

ELIGIBILITY:
Inclusion Criteria:

* Age between 25 and 65 years
* Continuous or recurrent episodes of pain in the lower back lasting for more than 12 weeks (chronic)
* No specific cause for pain complaints
* No other pathologic complaints or immobility
* Sufficient auditory and visual communication skills and
* Sufficient knowledge of the Turkish language

Exclusion Criteria:

* Any chronic disorder that may prevent exercise,
* Personal history of neurologic or rheumatologic disease,
* Pregnant or lactating women,
* Patients with malignancy or a lumbar comorbidity
* Terminal or progressive disease and any other musculoskeletal condition
* Surgery in the last 6 months and
* Any type of treatment for low back pain within past 6 months

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-05-11 (Actual); Primary Completion 2016-06-01 (Actual); Study Completion 2016-06-01 (Actual)

PRIMARY OUTCOMES:
Revised Oswestry Disability Index | 1 month
  Disability

IPD SHARING:
Plan to Share IPD: No